CLINICAL TRIAL: NCT00584363
Title: Pancreatic and Gastrointestinal Tumor Registry and Tissue Collection (UAB/UMN SPORE in Pancreatic Cancer)
Brief Title: Pancreatic and Gastrointestinal Tumor Registry and Tissue Collection
Acronym: SPORE
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charles Mel Wilcox, MD, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F040514008; 2P50CA101955 (NIH)
Record Dates: First submitted 2007-12-24; First posted 2008-01-02 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Specimens are frozen and stored
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to collect pancreatic tissue, blood and urine from adults to study pancreatic abnormalities.

DETAILED DESCRIPTION:
The aim of the study is to standardize, collect and share pancreatic cancer related information, to be used for research purposes only by researchers from different participating institutions/centers.

ELIGIBILITY:
Inclusion Criteria:

* Person over 19 years of age, patient with a tissue-proven diagnosis of pancreatic cancer at the University of Alabama at Birmingham (UAB) University Hospital during the period, and cognitive ability to provide informed consent

Exclusion Criteria:

* Person not 19 or older and have not had a tissue-proven diagnosis of pancreatic cancer.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 19 years of age or older, pancreatic cancer patients at the University of Alabam at Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2004-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To diagnose Pancreatic Cancer | 5 years

SECONDARY OUTCOMES:
Preventing patient form being misdiagnosed | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Wilcox, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States